CLINICAL TRIAL: NCT00046176
Title: A Phase III, 48-Week, Open-Label, Randomized, Multicenter Study of the Safety and Efficacy of the Abacavir/Lamivudine Fixed-Dose Combination Tablet Administered QD Versus Abacavir + Lamivudine Administered BID in Combination With a PI or NNRTI in Antiretroviral Experienced Patients.
Brief Title: A HIV Study Of A Fixed-Dose Combination Tablet In Antiretroviral Experienced Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESS30008
Record Dates: First submitted 2002-09-20; First posted 2002-09-23 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Infection, Human Immunodeficiency Virus I; HIV Infection
Keywords: HIV-1 Abacavir Lamivudine Antiretroviral-experienced
MeSH Terms: conditions — Infections; HIV Infections | interventions — abacavir, lamivudine drug combination; abacavir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: abacavir/lamivudine
Drug: abacavir
Drug: lamivudine
  Other Names: abacavir; abacavir/lamivudine

SUMMARY:
This study is a 48-week study designed to evaluate the safety and efficacy of a fixed-dose combination tablet administered once-a-day versus the individual tablets administered twice-a-day within 3-drug combination regimens in ART (antiretroviral)-experienced HIV-1 infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving an initial antiretroviral therapy (ART) regimen composed of the drug abacavir (ABC) 300mg twice a day, plus the drug 3TC (lamivudine) 150mg twice a day in combination with either a protease inhibitor or non-nucleoside reductase inhibitor (NNRTI) for at least 24 weeks.
* NOTE: Subjects who have required a change in initial protease inhibitor (PI) or NNRTI therapy due to intolerance (not treatment failure) are eligible. Subject must be on a stable regimen of the second PI or NNRTI therapy for at least 6 months before enrollment in this study.
* Plasma HIV-1 RNA less than 400 copies/mL for at least 3 months immediately preceding the screening visit, and at screening.
* CD4+ cell count of at least 50 cells/mm3 at screening.
* Written informed consent to participate in the study before participation.
* Male or female (Females of child-bearing potential must have a negative serum pregnancy test at screening and agree to an acceptable method of contraception.)

Exclusion Criteria:

* History of a CDC Clinical Category C event requiring treatment (not including cutaneous Kaposi's sarcoma) within 45 days of the screening visit. Treatment for the acute event must have been completed at least 30 days before screening.
* Subject is enrolled in one or more investigational drug studies which may impact HIV RNA suppression.
* Subject is unable to complete the 48-week dosing period, evaluations and assessments.
* Subject is pregnant or breastfeeding.
* History of clinically relevant inflammation of the pancreas or hepatitis within 6 months prior to screening.
* Subject suffers from a serious medical condition, such as diabetes or heart problem.
* Pre-existing mental, physical, or substance abuse disorder.
* History of inflammatory bowel disease or malignancy, intestinal ischemia, malabsorption, or other gastrointestinal dysfunction.
* Abnormal laboratory results within 28 days before the first dose of study medication.
* Required treatment with radiation therapy or cytotoxic chemotherapeutic agents within 28 days before screening, or will need these during the study.
* Subject requires treatment with immunomodulating drugs such as systemic corticosteroids, interleukins, vaccines, or interferons within 28 days prior to screening, or subject has received an HIV-1 immunotherapeutic vaccine within 90 days prior to screening.
* Asthmatic subjects using inhaled corticosteroids are eligible for enrollment.
* Subject requires treatment with foscarnet, hydroxyurea or other agents with documented activity against HIV-1 in vitro within 28 days of screening.
* Subject has a history of allergy to any of the study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2002-08-26 (Actual); Primary Completion 2004-05-17 (Actual); Study Completion 2004-05-17 (Actual)

PRIMARY OUTCOMES:
Proportion of non-virologic failures through Week 48. Treatment-limiting adverse events over 48 weeks. | 48 weeks

SECONDARY OUTCOMES:
Viral load response at Week 24 and 48 T-cell count Disease progression Health outcomes Resistance | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (41):
- United States (37):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Somers Point, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Reading, Pennsylvania
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Hampton, Virginia
- GSK Investigational Site, San José, Costa Rica
- GSK Investigational Site, Panama City, Panama
- Puerto Rico (2):
  - GSK Investigational Site, Ponce
  - GSK Investigational Site, Rio Piedras

REFERENCES:
- [Result] ABACAVIR + LAMIVUDINE FIXED DOSE COMBINATION TABLET ONCE DAILY (QD) COMPARED WITH ABACAVIR (ABC) AND LAMIVUDINE (3TC) TWICE DAILY (BID) IN HIV-1 INFECTED SUBJECTS (ESS30008). Hill-Zabala, Christina E. PharmD 1, Sosa, Nestor MD 2, DeJesus, Edwin MD 3, Herrera, Gisella MD, Florance, Allison M. MS , Watson, Maria E. PhD , and Shaefer, Mark S. PharmD (144F), 2005 Annual Meeting of the American College of Clinical Pharmacy, San Francisco, CA; USA, 10/23/2005
- [Result] EFFICACY AND SAFETY OF A ONCE DAILY FIXED-DOSE COMBINATION OF ABACAVIR/LAMIVUDINE (ABC/3TC) [FDC ] VERSUS ABC TWICE DAILY AND 3TC ONCE DAILY AS SEPARATE ENTITIES [SE] IN ART-EXPERIENCED HIV-1 INFECTED SUBJECTS (CAL30001): 48 WEEK DATA. Clumeck, N., LaMarca, A., Fu, K., Gordon, D., Craig, C., Zhao, H., Paes, D., and Scott, T. (WePe6.3C13), 3rd International AIDS Society Conference on HIV Pathogenesis and Treatment, Rio de Janeiro; Brazil, 7/24/2005
- [Result] Sosa N, DeJesus E, Hill-Zabala C, et al. Abacavir + lamivudine (ABC/3TC) fixed-dose combination tablet once-daily compared with abacavir and lamivudine twice-daily in HIV-1-infected subjects over 48 weeks (ESS30008). 2th Conference on Retroviruses and Opportunistic Infections, Boston, MA, February 22-25, 2005. [poster 572]
- [Result] PATIENT SATISFACTION WITH ABACAVIR (ABC)-LAMIVUDINE (3TC) FIXED DOSE COMBINATION (FDC) TABLET ONCE DAILY (QD) COMPARED WITH ABC AND 3TC TWICE DAILY (BID) IN HIV-1 INFECTED PATIENTS (ESS30008). Hill-Zabala, Christina E. PharmD , Watson, Maria E. PhD , Sosa, Nestor MD , DeJesus, Edwin MD , and Florance, Allison M. MS (145E), 2005 Annual Meeting of the American College of Clinical Pharmacy, San Francisco, CA; USA, 10/23/2005
- [Result] Sosa N, Hill-Zabala C, Dejesus E, Herrera G, Florance A, Watson M, Vavro C, Shaefer M. Abacavir and lamivudine fixed-dose combination tablet once daily compared with abacavir and lamivudine twice daily in HIV-infected patients over 48 weeks (ESS30008, SEAL). J Acquir Immune Defic Syndr. 2005 Dec 1;40(4):422-7. doi: 10.1097/01.qai.0000184859.24071.bd. PMID 16280696
- [Result] Sosa N, DeJesus E, Hill-Zabala C, et al. Abacavir + lamivudine (ABC/3TC) fixed-dose combination tablet once-daily compared with abacavir and lamivudine twice-daily in HIV-1-infected subjects (ESS30008). 7th International Congress on Drug Therapy in HIV Infection, Glasgow, UK, November 14-18, 2004 . [poster P45]